CLINICAL TRIAL: NCT03555968
Title: Determining the Combined Effects of THC and Alcohol on Driving Performance
Brief Title: Effects of THC and Alcohol on Driving Performance
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistical issues
Sponsor: Lakehead University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2018502
Record Dates: First submitted 2018-05-18; First posted 2018-06-14 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Cannabis; Alcohol Drinking; Accident, Traffic
Keywords: THC; Alcohol; Driving; Dronabinol
MeSH Terms: conditions — Marijuana Abuse; Alcohol Drinking | interventions — Dronabinol; nabiximols; THC 5

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- THC 0 + BAC 0 (Placebo Comparator): Participants will receive 0mg of THC in combination with blood alcohol concentrations of .000%.
  Interventions: Drug: THC 0; Other: BAC 0
- THC 5 + BAC 0 (Experimental): Participants will receive 5mg of THC in combination with blood alcohol concentrations of .000%.
  Interventions: Drug: THC 5; Other: BAC 0
- THC 10 + BAC 0 (Experimental): Participants will receive 10mg of THC in combination with blood alcohol concentrations of .000%.
  Interventions: Drug: THC 10; Other: BAC 0
- THC 5 + BAC .025 (Experimental): Participants will receive 5mg of THC in combination with blood alcohol concentrations of .025%.
  Interventions: Drug: THC 5; Other: BAC .025
- THC 10 + BAC .025 (Experimental): Participants will receive 125 µg/kg of THC in combination with blood alcohol concentrations of .025%.
  Interventions: Drug: THC 5; Other: BAC .025
- THC 0 + BAC .049 (Experimental): Participants will receive 0 µg/kg of THC in combination with blood alcohol concentrations of .049%.
  Interventions: Drug: THC 0; Drug: THC 10; Other: BAC .025; Other: BAC .049
- THC 5 + BAC .049 (Experimental): Participants will receive 5mg of THC in combination with blood alcohol concentrations of .049%.
  Interventions: Drug: THC 5; Other: BAC .049
- THC 10 + BAC .049 (Experimental): Participants will receive 10mg of THC in combination with blood alcohol concentrations of .049%.
  Interventions: Drug: THC 5; Other: BAC .049
- THC 0 + BAC .025 (Experimental): Participants will receive 0 µg/kg of THC in combination with blood alcohol concentrations of .025%.
  Interventions: Drug: THC 0; Drug: THC 10; Other: BAC .025; Other: BAC .049

INTERVENTIONS:
Drug: THC 0 — THC dose = 0mg
  Other Names: Tetrahydrocannabinol; Dronabinol; Cannabis
  Arms: THC 0 + BAC .025; THC 0 + BAC .049; THC 0 + BAC 0
Drug: THC 5 — THC dose = 5mg
  Other Names: Tetrahydrocannabinol; Dronabinol; Cannabis
  Arms: THC 10 + BAC .025; THC 10 + BAC .049; THC 5 + BAC .025; THC 5 + BAC .049; THC 5 + BAC 0
Drug: THC 10 — THC dose = 10mg
  Other Names: Tetrahydrocannabinol; Dronabinol; Cannabis
  Arms: THC 0 + BAC .025; THC 0 + BAC .049; THC 10 + BAC 0
Other: BAC 0 — Blood alcohol concentration = .000%
  Arms: THC 0 + BAC 0; THC 10 + BAC 0; THC 5 + BAC 0
Other: BAC .025 — Blood alcohol concentration = .025%
  Arms: THC 0 + BAC .025; THC 0 + BAC .049; THC 10 + BAC .025; THC 5 + BAC .025
Other: BAC .049 — Blood alcohol concentration = .049%
  Arms: THC 0 + BAC .025; THC 0 + BAC .049; THC 10 + BAC .049; THC 5 + BAC .049

SUMMARY:
Low blood concentrations of THC and alcohol appear to have a minimal effect on driving performance.However, there is a gap in the literature about the combined effects of THC and alcohol. There is little empirical evidence to determine whether the combination of THC and alcohol could be additive or multiplicative. This issue is particularly important when dealing with concentrations that are just below legal thresholds - it is important to identify if someone who may have consumed cannabis and alcohol, in quantities that do not exceed legal thresholds, may nonetheless be impaired to drive. Answering this question requires more research on the combined effects of THC and alcohol under tightly controlled experimental conditions. Hence, the purpose of this study is to determine the additive (or multiplicative) effect of standardized low doses of cannabis, in combination with low-doses of alcohol, on a number of outcome measures related to driving. The investigators will focus specifically on the effect of low blood concentrations of THC (0, 125, and 250 µg/kg) alone and in combination with low blood concentrations of alcohol (BAC 0%, .025%, and .049%). They shall determine the combined effect of THC and alcohol on physiological, cognitive, subjective measures of impairment, and simulated driving. This study will focus on younger adults because they have higher impaired driving rates than other age groups. As a secondary aim of the study, the investigators will examine whether previous driving and drug use history are correlated with driving decisions during the simulated drive and subjective measures. This study will contribute to the evidence base informing legislation, policy making, and law enforcement. This study is particularly timely given upcoming changes in legislation about cannabis, and because the combination of THC and alcohol, even below legal thresholds, may lead to impaired driving and crashes.

ELIGIBILITY:
Inclusion Criteria:

* BMI >18 and <30
* valid G2 or G Ontario driver's license
* live on-campus or within 15 minutes drive of campus
* speak fluent English

Exclusion Criteria:

* history of cardiovascular or psychiatric disorders
* current use of psychoactive medication
* current drug or alcohol abuse problem
* positive drug screen
* BAC level > .000%

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Demerit Points on Simulated Road Test | @2.5 hours
  Demerit points incurred for driving errors during a simulated a G2 exit exam (the final step in Ontario's graduated licensing framework) on a STISIM Drive 3-screen driving simulator; demerit points will be assigned in real-time by a member of the research team based on the Ontario Ministry of Transportation scoring scheme

SECONDARY OUTCOMES:
Standard Deviation of Lane Position in Meters (STISIM Drive-Recorded Variable) | @2.5 hours
  Recorded by the STISIM simulator during the simulation
Mean and Standard Deviation of Velocity in Meters/Second (STISIM Drive-Recorded Variable) | @2.5 hours
  Recorded by the STISIM simulator during the simulation
Mean and Standard Deviation of Acceleration in Meters/Second (STISIM Drive-Recorded Variable) | @2.5 hours
  Recorded by the STISIM simulator during the simulation
Blood Pressure (Systolic/Diastolic mmHg) | @25 minutes and 2 hours
  Systolic & diastolic blood pressure via automated blood pressure cuff
Heart Rate (BPM) & Heart Rate Variability via ECG | Hour 0-3.5
  Continuous heart rate in beats per minute via 3-lead electrocardiography recording; will allow for calculation of heart rate variability)
Electrical Brain Activity via EEG | Hour 0-3.5
  Continuous brain activity via electroencephalography recording
Median Response Time and Efficiency in Alerting, Orienting & Executive Attention as Measured by the Attention Network Test (in milliseconds) | @25 minutes and 2 hours
  A computerized test to measure participants' performance in three separate components of attention: alerting, orienting, and executive attention
Perceptual Motor Speed & Efficiency as Measured by Time (in seconds) to Complete Trail Making Tests A&B | @25 minutes and 2 hours
  A pen and paper test to measure perceptual motor speed and efficiency
Visual Analogue Scale of Perceived Effects | @25 minutes and 2 hours
  Ratings of participants' current perceptions of mood and bodily sensations (22 items including anxiety, alertness, dizziness, dry mouth) driving (3 items related to current willingness to drive), and subjective impairment (at time 2 only; 6 items related to strength of effects, perceived performance on tests); all items measures from not at all>extremely or absent>severe on a 100 mm line

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bédard, PhD, Principal Investigator — Lakehead University

IPD SHARING:
Plan to Share IPD: No